CLINICAL TRIAL: NCT01613833
Title: Evaluation of Serum and Synovium Protease Inhibitor Levels in Primary and Secondary Osteoarthritic Joints, and Comparison for Patients Undergoing Joint Replacement
Brief Title: Serum and Synovium Protease Inhibitor Levels in Primary and Secondary Osteoarthritic Joints
Status: Suspended | Type: Observational
Why Stopped: need new PI, i moved
Sponsor: Scuderi, Gaetano J., M.D. (Other)
Responsible Party: Sponsor
Other Study IDs: Scu.Cyt.003
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis of the Knee
Keywords: Alpha2 macroglobulin; Osteoarthritis; plasma and synovium
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Blood Specimen Collection; Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. 2cc whole blood to be collected from patient on date of total knee arthroplasty
  2. Joint aspirate harvested and collected intraoperatively during total knee arhtroplasty
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary OA Group: Subjects who are to undergo primary total knee arthroplasty due to primary OA which may include but is not limited to bilateral or peripheral involvement with no significant history of overuse or trauma to the joint.
  Interventions: Procedure: Blood Draw; Procedure: Joint Aspirate Harvest
- Secondary/Post-traumatic OA Group: Subjects who are to undergo primary total knee arthroplasty due to osteoarthritis of the knee that is secondary to injury or overuse of the joint.
  Interventions: Procedure: Blood Draw; Procedure: Joint Aspirate Harvest

INTERVENTIONS:
Procedure: Blood Draw — Blood drawn for A2M levels to be assayed at Cytonics
  Other Names: Phlebotomy
  Groups: Primary OA Group
Procedure: Joint Aspirate Harvest — Joint aspirate harvested for A2M levels to be assayed at Cytonics
  Other Names: Synoviual Fluid
  Groups: Primary OA Group
Procedure: Blood Draw — Blood drawn for A2M levels to be assayed at Cytonics
  Other Names: Phlebotomy
  Groups: Secondary/Post-traumatic OA Group
Procedure: Joint Aspirate Harvest — Joint aspirate harvested for A2M levels to be assayed at Cytonics
  Other Names: Synovial Fluid
  Groups: Secondary/Post-traumatic OA Group

SUMMARY:
Osteoarthritis (OA) is the irreversible degeneration of articular cartilage and underlying bone. It poses a major healthcare problem as it is the leading cause of joint disease and disability in the United States. It was traditionally thought that OA was a consequence of aging and joint trauma. However, it is now thought that OA is a result of the interplay of multiple genetic, biomechanical, and biochemical factors that disrupt the normal homeostasis of cartilage, bone, and synovium.

OA is classified into two groups, primary and secondary. Primary OA is classically polyarticular and peripheral while secondary OA can commonly be attributed to a specific cause, limited to a singular joint, and a result of trauma. It is known as post-traumatic OA (PTOA). Other causes of secondary OA include congenital disorders, calcium pyrophosphate dehydrate deposition disease, and other diseases. Regardless of classification, genetic variation in the normal metabolism of cartilage and bone is thought to play a role in the progression of OA. Furthermore, the polyarticular presentation of primary idiopathic osteoarthritis suggests that it may have a stronger genetic component as compared to secondary OA, indicating a deviation from normal cartilage and bone homeostasis.

Matrix metalloproteinases (MMP) and their inhibitors take part in the metabolism of cartilage and bone. MMPs are enzymes that catalyze the degradation of elements within joint spaces while their inhibitors cease this activity. Alpha-2-Macroglobulin (A2M) is a naturally-occurring plasma glycoprotein that functions throughout multiple tissues and extracellular spaces as a protease inhibitor but does not normally reach high levels within the intra-articular joint space. A2M is believed to modulate the systemic inflammatory response by its ability to bait, trap, and clear various MMPs and cytokines. Concentrated A2M directly addresses the roles of cytokines and catabolic enzymes known to participate in the development of osteoarthritis. Cytonics has shown that A2M can inhibit cartilage degradation in vitro. As the role of MMPs and protease inhibitors have emerged as key components of OA, the investigation of regulators of MMP has become of interest to elucidate the pathogenesis and possible novel treatments of OA.

This study aims to measure and correlate the levels of alpha-2-Macroglobulin (A2M) in plasma and knee joint OA between primary post-traumatic (PTOA) and secondary osteoarthritis groups.

DETAILED DESCRIPTION:
This is a single institution observational study.

Pre-procedure diagnosis: Based on chart review and consultation with operating surgeon of subjects undergoing total knee arthroplasty, patients will be grouped into primary or secondary (PTOA) osteoarthritis groups. Primary osteoarthritis will be identified through a clinical presentation of generalized osteoarthritis with possible bilateral involvement and no identifiable trauma or overuse to knee joint. Secondary osteoarthritis will be identified by history of overuse or trauma to the afflicted knee and a clinical presentation that in general lacks symmetrical involvement and/or severity, PTOA.

On the date of surgery, both primary and secondary groups will have 2 cc whole blood collected via venipuncture during placement of intravenous access for anesthesia. No additional venipuncture is necessary and this study necessitates no instrumentation/manipulation of patient beyond that of IV access normally obtained preoperatively. Blood will then be placed in refrigerated storage (2-6 C) until analyzed for A2M assay.

On the date of surgery, joint aspirate from both primary and secondary groups will be collected by the operating surgeon during knee arthroplasty. At the time of arthrotomy, joint fluid that is expressed from surgical site will be harvested and placed into an eppendorf tube and placed on ice. The study incurs no further risk to the patient and no further instrumentation/manipulation for synovial fluid harvest that is beyond the risk or instrumentation/manipulation of the indicated surgical procedure. Joint aspirates will then be stored until A2M assay.

ELIGIBILITY:
Inclusion Criteria:

Group 1, Non-traumatic primary OA:

1. Subject scheduled to undergo primary unilateral total knee arthroplasty for primary osteoarthritis as determined by an orthopedic surgeon
2. Subject is male or female over 45-75 years of age
3. Subject is able to read and understand informed consent form and must subsequently sign and date consent form

Group 2, Secondary post-traumatic/overuse OA:

1. Subject scheduled to undergo unilateral total knee arthroplasty secondary osteoarthritis as determined by an orthopedic surgeon, which MUST include either previous injury or surgery to the operative knee.
2. Subject is male or female 45-75 years of age
3. Subject is able to read and understand informed consent form and must subsequently sign and date consent form

Exclusion Criteria:

Group 1, Non-traumatic primary OA:

1. History of inflammatory arthritis (e.g. rheumatoid arthritis, ankylosing spondylitis)
2. Indication for surgery other than osteoarthritis
3. Revision total knee arthroplasty
4. Age >75, age <44
5. Unable to read, understand, or sign informed consent form
6. Previous knee infection
7. Congenital disorders of the knee, calcium pyrophosphate dehydrate deposition disease

Group 2, Secondary post-traumatic/overuse OA:

1. History of inflammatory arthritis (e.g. rheumatoid arthritis, ankyolosing spondylitis)
2. Indication for surgery other than osteoarthritis
3. Age >75, age <44
4. Unable to read, understand, or sign informed consent form
5. Previous knee infection
6. Congenital disorders of the knee, calcium pyrophosphate dehydrate deposition disease

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
A2M levels in plasma and synovium | Analyzed at the end of data collection within; approximately within 3 months of collection
  A2M levels will be drawn from plasma and synovium on the date of surgery for total knee arthroplasty. samples will then be stored properly and analyzed once data collection is complete.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Scuderi, MD, Principal Investigator — Stanford University, Dept. of Orthopedic Surgery
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

REFERENCES:
- [Background] Creamer P, Hochberg MC. Osteoarthritis. Lancet. 1997 Aug 16;350(9076):503-8. doi: 10.1016/S0140-6736(97)07226-7. No abstract available. PMID 9274595
- [Background] Heliovaara M, Makela M, Impivaara O, Knekt P, Aromaa A, Sievers K. Association of overweight, trauma and workload with coxarthrosis. A health survey of 7,217 persons. Acta Orthop Scand. 1993 Oct;64(5):513-8. doi: 10.3109/17453679308993681. PMID 8237314
- [Background] Spector TD, Hart DJ, Doyle DV. Incidence and progression of osteoarthritis in women with unilateral knee disease in the general population: the effect of obesity. Ann Rheum Dis. 1994 Sep;53(9):565-8. doi: 10.1136/ard.53.9.565. PMID 7979593
- [Background] Jordan JM, Luta G, Renner JB, Linder GF, Dragomir A, Hochberg MC, Fryer JG. Self-reported functional status in osteoarthritis of the knee in a rural southern community: the role of sociodemographic factors, obesity, and knee pain. Arthritis Care Res. 1996 Aug;9(4):273-8. doi: 10.1002/1529-0131(199608)9:43.0.co;2-f. PMID 8997916
- [Background] Woessner JF Jr. The family of matrix metalloproteinases. Ann N Y Acad Sci. 1994 Sep 6;732:11-21. doi: 10.1111/j.1749-6632.1994.tb24720.x. No abstract available. PMID 7978784
- [Background] Tchetverikov I, Lohmander LS, Verzijl N, Huizinga TW, TeKoppele JM, Hanemaaijer R, DeGroot J. MMP protein and activity levels in synovial fluid from patients with joint injury, inflammatory arthritis, and osteoarthritis. Ann Rheum Dis. 2005 May;64(5):694-8. doi: 10.1136/ard.2004.022434. PMID 15834054
- [Background] Luan Y, Kong L, Howell DR, Ilalov K, Fajardo M, Bai XH, Di Cesare PE, Goldring MB, Abramson SB, Liu CJ. Inhibition of ADAMTS-7 and ADAMTS-12 degradation of cartilage oligomeric matrix protein by alpha-2-macroglobulin. Osteoarthritis Cartilage. 2008 Nov;16(11):1413-20. doi: 10.1016/j.joca.2008.03.017. Epub 2008 May 15. PMID 18485748
- [Background] Murphy G, Nagase H. Reappraising metalloproteinases in rheumatoid arthritis and osteoarthritis: destruction or repair? Nat Clin Pract Rheumatol. 2008 Mar;4(3):128-35. doi: 10.1038/ncprheum0727. PMID 18253109